CLINICAL TRIAL: NCT04983576
Title: Risk Factors for Mechanical Failure After Spinal Fusion : an Observational Study
Acronym: RachideMDS
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Vincenzo Peccerillo, Physiotherapist Vincenzo Peccerilo, Istituto Ortopedico Rizzoli
Other Study IDs: CE-AVEC 354/2021/Oss/IOR
Record Dates: First submitted 2021-07-03; First posted 2021-07-30 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Spinal Fusion; Surgery--Complications; Spine Disease
MeSH Terms: conditions — Spinal Diseases | interventions — Spinal Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: spinal fusion — patients undergoing spinal fusion

SUMMARY:
The aim of this of study is to identify the incidence of mechanical failures after spinal fusion within one year of surgery and to assess the related risk factors.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing spine fusion and followed up for clinical checks in the year following the surgery .

Exclusion Criteria:

* patients undergoing spine surgery without the application of instrumentation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoind spine surgery with arthrodesis
Sampling Method: Probability Sample
Enrollment: 393 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
incidence of mechanical failure | up to 1 year from the surgery
  number of mechanical failure / total number of spinal fusion performed

SECONDARY OUTCOMES:
deambulation performed during hospitalization | up to the first day(up to 1 day) for ambulation from the surgery
  number of patients that are able to achieve ambulation after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Vincenzo Peccerillo, Bologna, BO, Italy